CLINICAL TRIAL: NCT00472433
Title: A Phase II Study of Alemtuzumab in Autoimmune Cytopenias
Brief Title: The Efficacy and Safety of Alemtuzumab in Auotoimmune Cytopenias
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: no eligible patient
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Collaborators: Bayer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH011003
Record Dates: First submitted 2007-04-25; First posted 2007-05-11 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Autoimmune Cytopenias
Keywords: Alemtuzumab in autoimmune cytopenias
MeSH Terms: interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alemtuzumab

SUMMARY:
The majority of cases of autoimmune cytopenias, which includes immune thrombocytopenia (ITP), autoimmune hemolytic anemia, autoimmune neutropenia (AIN) and pure red cell aplasia, will respond to conventional immunosuppressive therapy with or without splenectomy. There is, however, a group of patients with refractory or chronically relapsing autoimmune cytopenias causing life-threatening hemorrhages, infections or anemia. Further problems include the short- and long-term side-effects of corticosteroids, and the potential toxicity of immunosuppressive and cytotoxic agents. An alternative and less toxic approach in these patients may be the treatment with Campath-1H, a humanized IgG monoclonal antibody specific for the CD52 antigen and present on human lymphocytes and monocytes. The main effect of Campath-1H is on T cell and it results in a prolonged and profound depletion of the CD4 and CD8 subpopulations, particularly the CD4 population, and this might "reset" the immune system without the need for total immune ablation.Therefore, this study is designed to investigate safety and efficacy of repeated Campath treatment cycles in autoimmune cytopenia.In order to minimize possible side effects of accumulating Campath, the 3 treatment cycles will be administered in consecutively reduced doses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of the following autoimmune cytopenias:

   immune thromobocytopenia purpura (ITP) autoimmune hemolytic anemia (AIHA) autoimmune neutropenia (AIN) pure red cell aplasia (PRCA) and
2. Patients must have refractory disease according to the following criteria

   1. not respond to steroids or
   2. need prednisolone more than 15 mg/d for maintenance therapy
3. Complete work up for baseline evaluation and measurement
4. Age > 18 years
5. Patient's free written inform consent

Exclusion Criteria:

1. Patients with a known hypersensitivity to murine proteins or to any component of alemtuzumab
2. Patients with poor performance status (ECOG criteria of 3-4)
3. Serologic evidence of human immunodeficiency virus exposure
4. Patients with active uncontrolled infection. Patients that are HIV positive or test positive on HBs or HCV antigens.
5. Pregnant or lactating women
6. Serious medical or psychiatric illness which prevent informed consent
7. Patients who are likely to lost to follow up (eg, unwilling or difficult to return, cannot be contacted)
8. Patients with active malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To investigate the efficacy of alemtuzumab in terms of objective response rate (ORR: complete remission [CR], partial remission [PR]), progression free survival (PFS), and relapse rate in patients with autoimmune cytopenias

SECONDARY OUTCOMES:
To determine the safety profiles of alemtuzumab in patients with autoimmune cytopenias.

CONTACTS AND LOCATIONS:
Overall Officials: Wichean Mongkonsritragoon, M.D., Principal Investigator — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Phramongkutklao Hospital, Bangkok, Thailand